CLINICAL TRIAL: NCT06314191
Title: Comparative Study to Identify Biomarkers of Visceral Adipose Tissue Responsible for Symptomatic Gonarthrosis in Obese Patients
Brief Title: Adipose Tissue and Symptomatic Gonarthrosis
Acronym: TAGS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-AOIP-02
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Gonarthrosis; Obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthrose group (Experimental)
  Interventions: Other: blood sampling; Other: knee radiography
- controle group (Active Comparator)
  Interventions: Other: blood sampling; Other: knee radiography

INTERVENTIONS:
Other: blood sampling — blood sampling with analyses
Other: knee radiography — radiography of both knees in Schuss

SUMMARY:
1. Prevalence of osteoarthritis in France Osteoarthritis (OA) is a very common disease, affecting almost 15% of the population. It is responsible for a significant socio-economic cost in connection with the chronic and disabling pain it causes . Gonarthrosis is the most frequently encountered arthritic localization . In a large 2010 meta-analysis, the main risk factors for developing knee OA were shown to be obesity, previous knee trauma, hand OA, female gender and advanced age. Smoking appeared to have a moderate protective effect . The risk of developing gonarthrosis in obese patients is 2.6 times higher than in the general population. Hypercholesterolemia itself is a risk factor for osteoarthritis, as are increased plasma levels of specific fatty acids and lipoproteins Inflammatory mechanism in osteoarthritis. Studies have shown that plasma levels of C-reactive protein, can be used to estimate individual susceptibility to developing osteoarthritis over a lifetime . In osteoarthritis patients, plasma concentrations of TNF-α, IL-6 and IL-1 are abnormally high, which appears to contribute to cartilage loss in these subjects .

3. Inflammatory mechanism in obesity. Obesity induces systemic and local joint mechanical stresses that increase the risk of developing gonarthrosis in obese or overweight individuals . Beyond the simple mechanical aspect, a body of evidence supports the assertion that obesity is responsible for a systemic inflammatory state, deleterious to joints. 1) Obesity is associated with radiographic and symptomatic osteoarthritis in non-weight-bearing joints, such as the hand In overweight and obese adults, plasma levels of tumor necrosis factor alpha (TNF-α) and interleukin-6 (IL-6) are significantly increased .

3)Weight loss in obese subjects with osteoarthritis alleviates joint symptoms through reduced mechanical stress but also through reduced production and response of inflammatory products .

4. Common inflammatory mechanisms between adipose tissue and obesity. The relationship between adipose tissue and inflammation is complex given the different types of adipose tissue and the action of cells derived from it. Adipose tissue is an active endocrine organ composed of mature and developing adipocytes, as well as fibroblasts, endothelial cells and a wide range of immune cells, namely adipose tissue macrophages, neutrophils, eosinophils, mast cells, T cells and B cells. Adipose tissue is recognized as an endocrine organ that secretes a large number of inflammatory mediators, including cytokines (IL-1, IL-6, IL-8, TNF-α) and adipokines (leptin, adiponectin, resistin, visfatin). Communication between adipocytes and immune cells maintains tissue homeostasis. Obesity, however, can upset this balance.

Lipid metabolism and joint disorders have been shown to be linked . A high-fat diet may contribute to the development of osteoarthritis .

White and brown adipose tissue appear to play a complementary role in the development of osteoarthritis. Increased white adipose tissue in obesity is thought to create a systemic environment of increased inflammation through the release of pro-inflammatory cytokines and adipokines such as leptin and visfatin, all of which have been associated with osteoarthritis . Locally, white adipocytes in infra patellar adipose tissue are architecturally different in patients without gonarthrosis compared with those with knee osteoarthritis. This difference suggests that adipocyte gene expression is directly influenced by inflammation . In obese individuals, there is elevated IL-6 production in brown adipose tissue . Furthermore, it would appear that brown adipose tissue, unlike white, down-regulates the inflammatory profile of macrophages .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 30 and 55.
* Patient with BMI > 40 or Patient with BMI between 35-40 and presence of hypertension and/or diabetes and/or obstructive sleep apnea syndrome.
* Patients scheduled for bypass or SLEEVE bariatric surgery.
* Patients with symptomatic gonarthrosis or patients with no signs of osteoarthritis.
* Patients who have given written consent following written and oral information.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient having undergone knee ligamentoplasty.
* Patient with knee infiltration less than three months old.
* In the group of patients with no osteoarthritis, no known osteoarthritis or signs of osteoarthritis in a joint other than the knee.
* Patients treated with lipid-lowering or cholesterol-lowering drugs
* Postmenopausal patients
* Patient with weight change of more than 5% in the last 3 months
* Patients with known systemic inflammatory or autoimmune diseases
* Patients on special diets in the last 3 months (gluten-free, high-protein, low-carbohydrate diets)
* Patient with knee pain of secondary origin: tumor, inflammation, infection, fracture
* Patient with a contraindication to bariatric surgery
* Patient protected by law under guardianship or curatorship, or unable to participate in a clinical study under article L. 1121-16 of the French Public Health Code.
* Patient with insufficient command of the French language (assessed during interview).

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
lipolytic activity | baseline and perioperatively
  glycerol dosage in mg/dL
lipolysis measurement | baseline and perioperatively
  HSL dosage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No